CLINICAL TRIAL: NCT04347876
Title: Outcome of COVID-19 Cases Admitted to Hospital and ICU With Positive Tuberculin Test: Can Previous BCG Alter the Prognosis?
Brief Title: Outcome of COVID-19 Cases Based on Tuberculin Test: Can Previous BCG Alter the Prognosis?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU12
Record Dates: First submitted 2020-04-14; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; BCG Vaccination
Keywords: Outcome; COVID-19 pneumonia; BCG; Tuberculin test positive; Egypt
MeSH Terms: conditions — COVID-19 | interventions — Tuberculin Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: COVID-19 positive with positive tuberculin test
  Interventions: Diagnostic Test: Tuberculin test
- Group B: COVID-19 positive with negative tuberculin test
  Interventions: Diagnostic Test: Tuberculin test

INTERVENTIONS:
Diagnostic Test: Tuberculin test — Test the delayed hypersensitivity reaction and immunity to previous BCG vaccination

SUMMARY:
There is no evidence that the Bacille Calmette-Guérin vaccine (BCG) protects people against infection with COVID-19 virus. Two clinical trials addressing this question are underway, and WHO will evaluate the evidence when it is available. In the absence of evidence, WHO does not recommend BCG vaccination for the prevention of COVID-19. WHO continues to recommend neonatal BCG vaccination in countries or settings with a high incidence of tuberculosis. There is experimental evidence from both animal and human studies that the BCG vaccine has non-specific effects on the immune system. These effects have not been well characterized and their clinical relevance is unknown

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive cases admitted to hospitals in Upper Egypt

Exclusion Criteria:

* None

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases admitted with proven COVID-19 positive disease will be included, tested with tuberculin test positive and negative ( History of previous BCG or not)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-06-16 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Pneumonia severity index | 2 weeks
  severity of COVID-19 pneumonia
Need for ICU admission | 2 weeks
  severe pneumonia indicating invasive or non invasive mechanical ventilation

SECONDARY OUTCOMES:
COVID -19 test conversion | 2 weeks
  number of days to cure from COVID-19 disease
Mortality | 2 weeks
  frequency of fatalities

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided